CLINICAL TRIAL: NCT04365426
Title: Effects of Oral Contraceptives on Diffuse Noxious Inhibitory Stimulus (DNIC) in Non-painful Healthy Women
Brief Title: Effects of Oral Contraceptives on DNIC in Non-painful Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Vina del Mar (Other)
Responsible Party: Principal Investigator, Nicolás Pinto Pardo, DDS, Msc, Ph.D, Universidad Vina del Mar
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Contraceptive Usage; Diffuse Noxious Inhibitory Control
MeSH Terms: conditions — Contraception Behavior | interventions — Cold Temperature; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral contraceptive (OC) (Experimental): Oral contraceptive patients will be tested to mechanical (cephalic and extracephalic) stimulus and cold pain stimulus.
  Interventions: Device: Mechanical stimulus; Procedure: Thermal (cold) stimulus; Other: Oral contraceptive (OC)
- No oral contraceptive (No OC) (Experimental): No oral contraceptive patients will be tested to mechanical (cephalic and extracephalic) stimulus and cold pain stimulus.
  Interventions: Device: Mechanical stimulus; Procedure: Thermal (cold) stimulus; Other: No oral contraceptive (No OC)

INTERVENTIONS:
Device: Mechanical stimulus — Electrical dynamometer to measure mechanical pressure
Procedure: Thermal (cold) stimulus — Water cold bath
Other: Oral contraceptive (OC) — Oral contraceptive (OC)
  Arms: Oral contraceptive (OC)
Other: No oral contraceptive (No OC) — No oral contraceptive (No OC)
  Arms: No oral contraceptive (No OC)

SUMMARY:
The purpose of this study is tu assess the influence of oral contraceptives (OC) on diffuse noxious inhibitory control (DNIC) in healthy women, tested during high, low endogenous estrogens sessions and ovulatory period.

DETAILED DESCRIPTION:
After being informed about the study and it protocol, all patients giving written informed consent, will undergo to a cephalic (masseter) and extracephalic (finger) mechanical stimulus to evaluate the threshold of mechanical pain, and physiological records of systolic/diastolic pressure and heart rates. After, we will evaluate the threshold response and physiological rates to the same mechanical stimulus under a thermal (cold) conditional pain (TCP) at 3 different moments of menstrual period in No contraceptive group (No OC) versus Contraceptive group (CO). Finally, we will compare the mechanical threshold response, physiological rates and pain perception between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women with oral contraceptive treatment (for at least 3 consecutive months), greater than or equal to 15 years old.
* Healthy women without oral contraceptive treatment, greater than or equal to 15 years old.
* Non pregnant women.
* Not under convulsive, chronic pain, antidepresive, antihypertensive, pharmacological treatments
* Without systemic pathologies.

Exclusion Criteria:

* Treatment of a pain, depression, hypertension, convulsion condition with or without medication.
* Regular use of benzodiazepines.
* Systemic pathologies
* Pregnant women
* Menopausal women

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Diffuse Noxious Inhibitory Control Efficiency in oral contraceptive healthy women | Baseline phase 1 (2-5 days), phase 2 (14-17 days), and phase 3 (21-27 days) after the beginning of menstrual period
  The efficiency of diffuse noxious inhibitory control (DNIC) is a measure of one's ability to inhibit pain perception. DNIC efficiency is assessed by a psychophysical test that involves a mechanical pressure in the masseter (cephalic) and finger (extracephalic) stimulus as the "test stimulus" and a cold-water bath as the "conditioning stimulus". The results of this test will be used as the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolás Pinto-Pardo, DDS, Ms, Ph.D, Principal Investigator — Universidad Vina del Mar
Locations (1):
- Universidad Viña del Mar, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No